CLINICAL TRIAL: NCT00293267
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Antiretroviral Activity of MK-0518 in Combination With an Optimized Background Therapy (OBT), Versus Optimized Background Therapy Alone, in HIV-Infected Patients With Documented Resistance to at Least 1 Drug in Each of the 3 Classes of Licensed Oral Antiviral Therapies
Brief Title: A Study to Evaluate the Safety and Efficacy of Raltegravir (MK0518) in HIV-Infected Patients Failing Current Antiretroviral Therapies (MK0518-018 EXT2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-018; 2005_096
Record Dates: First submitted 2006-02-14; First posted 2006-02-17 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): raltegravir potassium
  Interventions: Drug: raltegravir potassium
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: raltegravir potassium — Raltegravir 400 mg twice daily (b.i.d.) by mouth (p.o.) with optimized background therapy. Treatment period of 48 weeks.
  Other Names: ISENTRESS™
  Arms: 1
Drug: Comparator: Placebo — Placebo b.i.d. p.o. with optimized background therapy. Treatment period of 48 weeks.
  Arms: 2

SUMMARY:
This study will investigate the safety and efficacy of raltegravir as a therapy for HIV-infected patients failing current therapy with 3-class antiviral resistance.

DETAILED DESCRIPTION:
The primary double-blind study of raltegravir versus placebo was extended to 156 weeks and was followed by an open-label raltegravir phase in which continuing participants from both the raltegravir and placebo groups received open-label raltegravir for an additional 84 weeks for a maximum duration of up to 240 weeks. Participants who had viral failure after Week 16 may have received open-label raltegravir until Week 240.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV positive with HIV RNA values that are within ranges required by the study
* Patient must have documented failure of certain antiretroviral therapy
* Patient must be on the same antiretroviral therapy for at least the past two months

Exclusion Criteria:

* Patient is less than 16 years old
* Additional study criteria will be discussed and identified by the study doctor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Steigbigel RT, Cooper DA, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Nguyen BY, Teppler H; BENCHMRK Study Teams. Raltegravir with optimized background therapy for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):339-54. doi: 10.1056/NEJMoa0708975. PMID 18650512
- [Background] Cooper DA, Steigbigel RT, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Teppler H, Nguyen BY; BENCHMRK Study Teams. Subgroup and resistance analyses of raltegravir for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):355-65. doi: 10.1056/NEJMoa0708978. PMID 18650513
- [Result] Steigbigel RT, Cooper DA, Teppler H, Eron JJ, Gatell JM, Kumar PN, Rockstroh JK, Schechter M, Katlama C, Markowitz M, Yeni P, Loutfy MR, Lazzarin A, Lennox JL, Clotet B, Zhao J, Wan H, Rhodes RR, Strohmaier KM, Barnard RJ, Isaacs RD, Nguyen BY; BENCHMRK Study Teamsa. Long-term efficacy and safety of Raltegravir combined with optimized background therapy in treatment-experienced patients with drug-resistant HIV infection: week 96 results of the BENCHMRK 1 and 2 Phase III trials. Clin Infect Dis. 2010 Feb 15;50(4):605-12. doi: 10.1086/650002. PMID 20085491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 3; First Patient In: Mar 2006; Last Patient Last Visit (LPLV) Week 48: Aug 2007; 61 of 63 sites in Australia, Belgium, Denmark, France, Germany, Italy, Peru, Portugal, Spain, Switzerland, Taiwan, Thailand randomized patients. Extension Study LPLV Week 240: June 2011
Pre-assignment Details: Patients failed prior antiretroviral therapy (HIV RNA >1000 copies/mL), and had documented resistance to at least one drug in each class of licensed oral antiretroviral therapy (Nucleoside Reverse Transcriptase inhibitors, Non-Nucleoside Reverse Transcriptase inhibitors and Protease Inhibitors). All patients must have met laboratory criteria.
Period: Primary Study - Double-Blind Week 0-48
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 234 | 118
Treated | 232 | 118
Continuing in Double-Blind | 193 (Excludes participants who entered the open-label post virological failure (OLPVF) phase) | 50
Completed | 193 | 50
Not Completed | 41 | 68
Not completed — Never Treated | 2 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Death | 3 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Entered OLPVF Phase | 33 | 60
Period: Extension - Double-Blind Week 49-156
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 191 (2 participants who completed Week 48 did not enter the extension study) | 50
Completed | 139 | 35
Not Completed | 52 | 15
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 7 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Death | 3 | 0
Not completed — Participant relocated or site terminated | 2 | 0
Not completed — Other Reason | 7 | 0
Not completed — Entered OLPVF Phase | 15 | 6
Period: Extension - Open-Label Week 157-240
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 131 (8 of 139 participants who completed the double-blind phase did not enter this open-label phase) | 28 (7 of 35 participants who completed the double-blind phase did not enter this open-label phase)
Completed | 111 | 26
Not Completed | 20 | 2
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 7 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Participant relocated or site terminated | 2 | 0
Not completed — Other Reason | 3 | 1
Period: Open-Label Post Virologic Failure Phase
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 48 (Number of participants who failed treatment and consented to enter the OLPVF phase) | 66 (Number of participants who failed treatment and consented to enter the OLPVF phase)
Completed | 15 | 29
Not Completed | 33 | 37
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 23 | 19
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Laboratory Adverse Event | 0 | 2
Not completed — Participant Moved or Site Terminated | 0 | 2
Not completed — Other Reason | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT | Total
Number analyzed (Participants) | 232 | 118 | 350
Age, Continuous [Mean (Full Range); unit: Years] | 46.1 [16 to 74] | 43.7 [19 to 64] | 45.3 [16 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 15 | 52
  Male | 195 | 103 | 298
Race/Ethnicity, Customized [Number; unit: participants]
  White | 174 | 96 | 270
  Black | 18 | 5 | 23
  Asian | 14 | 5 | 19
  Hispanic | 6 | 1 | 7
  Other | 20 | 11 | 31
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: cells/mm^3] | 156 [1 to 792] | 153 [3 to 759] | 155 [1 to 792]
Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) [Geometric Mean (Full Range); unit: copies/mL] | 40519 [441 to 750000] | 31828 [200 to 750000] | 37352 [200 to 750000]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving HIV RNA <400 Copies/mL at Week 16
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 16
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 117
Percentage of Participants | 77.7 [71.8 to 82.9] | 41.0 [32.0 to 50.5]

2. Secondary Outcome: Percentage of Participants Achieving HIV RNA <50 Copies/mL at Week 16
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 16
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 117
Percentage of Participants | 61.6 [54.9 to 67.9] | 33.3 [24.9 to 42.6]

3. Secondary Outcome: Percentage of Participants Achieving HIV RNA <50 Copies/mL at Week 48
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 48
Time Frame: 48 Weeks
Population: Participants who experienced virologic failure after Week 16 are also counted as treatment failures for the subsequent virologic efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 231 | 118
Percentage of Participants | 64.5 [58.0 to 70.7] | 31.4 [23.1 to 40.5]

4. Secondary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Achieving HIV RNA <50 Copies/mL
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 156
Time Frame: 156 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 232 | 117
Percentage of Participants | 53.4 [46.8 to 60.0] | 25.6 [18.0 to 34.5]

5. Secondary Outcome: Open-Label Extension - Week 240: Percentage of Participants Achieving HIV RNA <50 Copies/mL
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 240
Time Frame: 240 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Raltegravir 400 mg b.i.d. + OBT: Raltegravir 400 mg b.i.d plus OBT includes all participants initially randomized to raltegravir. Those who did not experience virologic failure by Week 156 may have continued into the open-label phase. During the open-label phase, these participants continued to receive raltegravir plus OBT until Week 240.
- Placebo + OBT: Placebo plus OBT includes all participants initially randomized to placebo. Those who did not experience virologic failure by Week 156 may have continued into the open-label phase. During the open-label phase, these participants received raltegravir plus OBT until Week 240.
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 232 | 118
Percentage of Participants | 42.2 [35.8 to 48.9] | 18.6 [12.1 to 26.9]

6. Primary Outcome: Percentage of Participants Achieving HIV RNA <400 Copies/mL at Week 48
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 48
Time Frame: 48 Weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 231 | 118
Percentage of Participants | 73.6 [67.4 to 79.2] | 36.4 [27.8 to 45.8]

7. Secondary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Without Loss of Virologic Response
Description: For participants with confirmed HIV RNA levels <50 copies/mL on 2 consecutive visits, loss of virologic response is the occurrence of the first value >50 copies/mL or loss to follow-up; participants who never achieved HIV RNA <50 copies/mL on 2 consecutive visits are also considered as having loss of virologic response. Events are the numbers of participants with loss of virologic response versus the numbers of participants with no loss of virologic response (event free).
Time Frame: 156 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 232 | 118
Percentage of Participants | 47.4 | 24.6

8. Secondary Outcome: Change From Baseline in HIV RNA (log10 Copies/mL) at Week 16
Description: Mean change from baseline at Week 16 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 16
Population: Observed mean change from baseline in log10 plasma HIV RNA calculated using conventional imputation (replace <400 copies by 400 copies if signal detected; 200 copies if not detected); Missing values: baseline carry-
  forward for all failures/discontinued due to lack of efficacy
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 231 | 118
HIV RNA (log10 copies/mL) | -1.85 [-1.97 to -1.73] | -0.78 [-0.97 to -0.59]

9. Secondary Outcome: Change From Baseline in HIV RNA (log10 Copies/mL) at Week 48
Description: Mean change from baseline at Week 48 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 48
Population: Observed mean change from baseline in log10 plasma HIV RNA calculated using conventional imputation (replace <400 copies by 400 copies if signal detected; 200 copies if not detected); Missing values: baseline carry-forward for all failures/discontinued due to lack of efficacy
  Participants with virologic failure after Week 16 = treatment failures
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 231 | 118
HIV RNA (log10 copies/mL) | -1.67 [-1.81 to -1.54] | -0.68 [-0.86 to -0.50]

10. Secondary Outcome: Double-Blind Extension - Week 156: Change From Baseline in HIV RNA (log10 Copies/mL)
Description: Mean change from baseline at Week 156 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 156
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 207 | 107
HIV RNA (log10 copies/mL) | -1.44 [-1.60 to -1.28] | -0.51 [-0.67 to -0.34]

11. Secondary Outcome: Open-Label Extension - Week 240: Change From Baseline in HIV RNA (log10 Copies/mL)
Description: Mean change from baseline at Week 240 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 240
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 188 | 100
HIV RNA (log10 copies/mL) | -1.24 [-1.42 to -1.07] | -0.45 [-0.62 to -0.27]

12. Primary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Achieving HIV RNA <400 Copies/mL
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 156
Time Frame: 156 Weeks
Population: The analysis population was based on a non-completer equals failure approach where missing values for participants who discontinued the study for any reason were considered treatment failures.
  Participants who experienced virologic failure after Week 16 are counted also as treatment failures for the subsequent virologic efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 232 | 117
Percentage of Participants | 57.3 [50.7 to 63.8] | 25.6 [18.0 to 34.5]

13. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at Week 16
Description: Mean change from baseline at Week 16 in CD4 Cell Count (cells/mm^3)
Time Frame: Baseline and Week 16
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 cell count (cells/mm^3) was carried forward for participants who discontinued assigned therapy due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 231 | 118
CD4 Cell Count (cells/mm^3) | 82.7 [70.5 to 94.9] | 31.3 [17.8 to 44.8]

14. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at Week 48
Description: Mean change from baseline at Week 48 in CD4 Cell Count (cells/mm^3)
Time Frame: Baseline and Week 48
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 cell count (cells/mm^3) was carried forward for participants who discontinued assigned therapy due to lack of efficacy.
  Participants with virologic failure after Week 16 are treatment failures for virologic efficacy analyses.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 230 | 119
CD4 Cell Count (cells/mm^3) | 120.2 [102.2 to 138.1] | 49.4 [30.4 to 68.5]

15. Primary Outcome: Open-Label Extension - Week 240: Percentage of Participants Achieving HIV RNA <400 Copies/mL
Description: Percentage of participants who achieved HIV RNA <400 Copies/mL at Week 240
Time Frame: 240 Weeks
Population: The analysis population was based on a non-completer equals failure approach where missing values for participants who discontinued the study for any reason were considered treatment failures.
  Participants who experienced virologic failure after Week 16 are also counted as treatment failures for the subsequent virologic efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 232 | 118
Percentage of Participants | 45.3 [38.7 to 51.9] | 20.3 [13.5 to 28.7]

16. Secondary Outcome: Double-Blind Extension - Week 156: Change From Baseline in CD4 Cell Count (Cells/mm^3)
Description: Mean change from baseline at Week 156 in CD4 Cell Count (cells/mm^3)
Time Frame: Baseline and Week 156
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 207 | 107
CD4 Cell Count (cells/mm^3) | 170.9 [144.4 to 197.4] | 71.03 [46.28 to 95.77]

17. Secondary Outcome: Open-Label Extension - Week 240: Change From Baseline in CD4 Cell Count (Cells/mm^3)
Description: Mean change from baseline at Week 240 in CD4 Cell Count (cells/mm^3)
Time Frame: Baseline and Week 240
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 186 | 101
CD4 Cell Count (cells/mm^3) | 193.6 [159.1 to 228.0] | 68.2 [38.2 to 98.2]

ADVERSE EVENTS:
Time Frame: 240 Weeks
Description: Adverse events are reported by original treatment group for the entire 240-week study, including double-blind, open-label, and OLPVF phases; 94 of 118 participants in the placebo group also received raltegravir in the open-label or OLPVF phase.
Groups:
- Raltegravir 400 mg b.i.d Plus OBT: Includes all participants initially randomized to raltegravir, including those without virologic failure who
  continued into the open-label phase at Week 156 and those who entered the OLPVF phase due to virologic failure. During either open-label phase up to Week 240, these participants continued to receive raltegravir 400 mg b.i.d. plus OBT.
- Placebo Plus OBT: Includes all participants initially randomized to placebo, including those without virologic failure who continued into the open-label phase at Week 156 and those who entered the OLPVF phase due to virologic failure. During either open-label phase up to Week 240, these participants continued to receive raltegravir 400 mg b.i.d. plus OBT.
Arm/Group | Raltegravir 400 mg b.i.d Plus OBT | Placebo Plus OBT
Serious Adverse Events (participants affected / at risk) | 97/232 | 46/118
Other Adverse Events (participants affected / at risk) | 206/232 | 104/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 400 mg b.i.d Plus OBT (N=232) | Placebo Plus OBT (N=118)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (5) | 2 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Myxoedema (Endocrine disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (11)
Soft tissue inflammation (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 2 (3) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Anogenital warts (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Choriomeningitis lymphocytic (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Disseminated cytomegaloviral infection (Infections and infestations) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 1 (1)
End stage AIDS (Infections and infestations) | 1 (1) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (2) | 0 (0)
Epidermodysplasia verruciformis (Infections and infestations) | 0 (0) | 1 (1)
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1)
Fallopian tube abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 3 (3) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (4)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 3 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 5 (6)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (3) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis of genitourinary system (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Visceral leishmaniasis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8) | 3 (3)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 3 (5)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 2 (3)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (4)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Disturbance in social behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Varicophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 400 mg b.i.d Plus OBT (N=232) | Placebo Plus OBT (N=118)
Anaemia (Blood and lymphatic system disorders) | 9 (12) | 7 (13)
Lymphadenopathy (Blood and lymphatic system disorders) | 19 (19) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 15 (16) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 74 (110) | 34 (70)
Gastritis (Gastrointestinal disorders) | 8 (8) | 7 (8)
Haemorrhoids (Gastrointestinal disorders) | 12 (12) | 2 (2)
Nausea (Gastrointestinal disorders) | 30 (38) | 20 (25)
Vomiting (Gastrointestinal disorders) | 18 (26) | 17 (25)
Asthenia (General disorders) | 15 (16) | 11 (11)
Fatigue (General disorders) | 18 (18) | 6 (9)
Injection site reaction (General disorders) | 18 (19) | 14 (16)
Pyrexia (General disorders) | 28 (35) | 18 (23)
Anogenital warts (Infections and infestations) | 11 (14) | 6 (7)
Bronchitis (Infections and infestations) | 42 (71) | 16 (23)
Gastroenteritis (Infections and infestations) | 22 (28) | 3 (4)
Genital herpes (Infections and infestations) | 10 (11) | 9 (12)
Herpes simplex (Infections and infestations) | 12 (13) | 3 (6)
Herpes zoster (Infections and infestations) | 20 (23) | 7 (10)
Influenza (Infections and infestations) | 25 (28) | 8 (11)
Nasopharyngitis (Infections and infestations) | 58 (96) | 21 (51)
Oral candidiasis (Infections and infestations) | 11 (14) | 15 (20)
Pharyngitis (Infections and infestations) | 15 (24) | 8 (11)
Pneumonia (Infections and infestations) | 9 (12) | 9 (11)
Respiratory tract infection (Infections and infestations) | 19 (21) | 3 (5)
Sinusitis (Infections and infestations) | 11 (15) | 6 (13)
Upper respiratory tract infection (Infections and infestations) | 20 (35) | 7 (15)
Urinary tract infection (Infections and infestations) | 14 (17) | 6 (8)
Alanine aminotransferase increased (Investigations) | 24 (40) | 9 (19)
Aspartate aminotransferase increased (Investigations) | 24 (30) | 8 (18)
Blood cholesterol increased (Investigations) | 28 (44) | 9 (20)
Blood triglycerides increased (Investigations) | 22 (30) | 11 (14)
Weight decreased (Investigations) | 6 (8) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 6 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (7) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (33) | 10 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (15) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16) | 6 (6)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (20) | 6 (8)
Dizziness (Nervous system disorders) | 14 (15) | 2 (2)
Headache (Nervous system disorders) | 28 (38) | 24 (29)
Depression (Psychiatric disorders) | 13 (14) | 9 (10)
Insomnia (Psychiatric disorders) | 24 (24) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 11 (14)
Eczema (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (7)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (20) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 20 (25) | 7 (12)
Hypertension (Vascular disorders) | 32 (32) | 12 (12)

LIMITATIONS AND CAVEATS:
Adverse events are reported by original treatment group for the entire 240-week study, including double-blind, open-label, and OLPVF phases; 94 of 118 participants in the placebo group also received raltegravir in the open-label or OLPVF phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.